CLINICAL TRIAL: NCT03601598
Title: A Phase Ib/II , Open-label , Investigator-initiated Trail of An Anti-PD-1 Inhibitor SHR-1210 in Combination With A CDK4/6 Inhibitor SHR6390 in Patients With Advanced Colorectal Cancer, Non-small Cell Lung Cancer and Hepatocellular Carcinoma
Brief Title: A Trial of SHR-1210 in Combination With SHR6390 in Patients With Advanced CRC, NSCLC and HCC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Harbin Medical University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yanqiao Zhang, Director of the hospital, Harbin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-SHR6390-IIT
Record Dates: First submitted 2018-07-13; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: CRC; HCC; NSCLC
MeSH Terms: interventions — camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1210 + SHR6390 (Experimental): SHR-1210 was administered 200mg iv every 2 weeks in combination with SHR6390 150mg or 100mg oral daily with 3 weeks on and 1 week off
  Interventions: Drug: SHR-1210; Drug: SHR6390

INTERVENTIONS:
Drug: SHR-1210 — SHR-1210 was administered 200mg iv every 2 weeks
Drug: SHR6390 — SHR6390 was administered 150mg or 100mg oral daily with 3 weeks on and 1 week off

SUMMARY:
This is a Phase Ib/II , Open-label , Investigator-initiated Trail of SHR-1210 (an Anti-PD-1 Inhibitor) in Combination With SHR6390 (a CDK4/6 Inhibitor) in Patients With Advanced Colorectal Cancer, Non-small Cell Lung Cancer and Hepatocellular Carcinoma.

The study was designed in two stages, the first stage was the tolerance observation stage, and the second stage was the curative effect expansion stage.

The first part of the study is the Dose-finding Phase designed to establish the safety of SHR-1210 Combination With SHR6390 at different dose Levels(150mg QD or 100mg QD ). The second part of the study is the Expansion Phase designed to generate additional clinical data at specified doses .

This study aims to evaluate the safety and efficacy of SHR-1210 combination with SHR6390 in the treatment of advanced CRC,NSCLC and HCC.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in this study and sign informed consent .
* Men or women aged 18-75 years
* Has confirmed by histology and cytology advanced and/or metastatic colorectal cancer patients, the advanced (Ⅲ B/Ⅳ period) in non-small cell lung cancer，Or patients with advanced hepatocellular carcinoma confirmed histologically or cytologically or clinically，At least one measurable lesion that meets the RECIST v1.1 criteria without local treatment.
* The patients can swallow pills normally.
* ECOG score was 0 or 1.
* Have a life expectancy of at least 12 weeks.
* The functions of vital organs meet the following requirements (excluding the use of any blood components and cytokines during screening) : Neutrophils≥1.5 x 109/L, Hb≥9g/dL; Plt≥90 x 109/L, ALB≥3g/dL, TSH≤ULN(Upper Limit Of Norma), TBIL ≤ 1.25 x ULN, ALT and AST ≤ 1.5 x ULN, AKP≤ 2.5 x ULN, CR≤ 1.5 x ULN
* Female Subjects of childbearing potential must have a negative serum pregnancy test within 72 hours before the first dose and must be willing to use very efficient barrier methods of contraception for the course of the study through 3 months after the last dose of study treatment.

Exclusion Criteria:

* Subjects had any active autoimmune disease or history of autoimmune disease.
* Subjects are using immunosuppressive agents, or systemic, or absorptive,local hormone therapy to achieve immunosuppression. It is still in use within 2 weeks before enrollment.
* Subjects with severe allergic reactions to other monoclonal antibodies.
* The subjects had a central nervous system metastases of clinical symptoms.
* Central lung squamous cell carcinoma, or NSCLC with large vascular invasion confirmed by imaging.
* A heart condition or disease that is not well controlled.
* Subjects had active infections.
* Other clinical trials of drugs were used within 4 weeks prior to the first administration.
* The subjects have received other PD-1 antibody therapy or other immunotherapy for PD-1 / PD-L1 or CDK4/6 inhibitor treatment in the past.
* There are other factors lead to patients can not participate in this clinical study by the judgment of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2018-07-30 (Estimated); Primary Completion 2019-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
MTD /DLT (phase Ib) | Within four weeks after dosing
  Maximum Tolerated Dose/Dose Limiting Toxicity
ORR(phase II) | from the first drug administration up to two years
  Overall Response Rate

SECONDARY OUTCOMES:
ORR(phase Ib) | from the first drug administration up to two years
  Overall Response Rate
Incidence of Treatment-Emergent Adverse Events (phase Ib/II) | from the first drug administration to within 90 days for the last SHR-1210 dose
  adverse events/serious adverse events
CBR (phase Ib/II) | from the first drug administration up to last patients treatment for 6 months.
  Clinical Benefit Rate
DoR (phase Ib/II) | from the first drug administration up to two years
  Duration of response
PFS(phase Ib/II) | from the first drug administration up to two years
  Progression-Free-Survival
TTR(phase Ib/II) | from the first drug administration up to one year
  Time to Response
12m-OS | 12 months after the first drug administration
  12 months Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Yanqiao Zhang, PhD, Principal Investigator — Harbin Medical University Cancer Hosptital